CLINICAL TRIAL: NCT04661696
Title: Efficacy and Safety of Paclitaxel (Albumin-bound) Combination With Carboplatin in the Treatment of Platinum-sensitive Recurrent Ovarian Cancer: a Multicenter, Open, Phase 2 Clinical Study
Brief Title: Efficacy and Safety of Paclitaxel (Albumin-bound) Combination With Carboplatin in Ovarian Cancer.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ling-Ying Wu, chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19/339-2123
Record Dates: First submitted 2020-11-30; First posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Taxes; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-arm (Experimental): Paclitaxel (albumin-bound) 130 mg/m2, i.v., d1, 8; Carboplatin AUC 5, i.v. d1; repeat every 21days, 6 cycles.
  Interventions: Drug: Paclitaxel (albumin-bound)

INTERVENTIONS:
Drug: Paclitaxel (albumin-bound) — The dose of intravenous chemotherapy drug is calculated according to the body surface area.When patients have serious adverse events, dose suspension and dose reduction are allowed. Paclitaxel (albumin-bound) was allowed to be reduced only twice (20% standard dose reduction in the first dose and 20% lower in the second dose).Once the dose is reduced, all subsequent doses should be maintained at reduced dosage.
  Other Names: carboplatin

SUMMARY:
Epithelial ovarian cancer is the most fatal gynecological malignancy. Despite initial therapeutic response, the majority of advanced-stage patients relapse and eventually succumb to chemoresistant disease. The majority of ovarian cancer patients with standardized treatment, including tumor cell reduction and postoperatively platinum-based combination chemotherapy, will still experience tumor recurrence and multiple recurrences within 6-18 months.With the increase in the number of recurrences, the intertherapeutic period will shorten and eventually drug resistance will emerge.The purpose of treatment for recurrent ovarian cancer is mainly to improve the quality of life of patients and prolong survival. CSPC OUYI PHARMACEUTICAL CO., LTD has successfully developed Paclitaxel (Albumin-Bound) and the bioequivalence test results show good consistency with Abraxane.To evaluate the efficacy and safety of Paclitaxel (Albumin-Bound) combination with carboplatin in Chinese patients with platinum-sensitive recurrent ovarian cancer, this clinical study is planned.

DETAILED DESCRIPTION:
This study is a multicenter, open, single arm, phase 2 clinical study in patients with platinum-sensitive recurrent ovarian cancer.75 patients were planned to be enrolled, and the eligible patients were given the following regimen: Paclitaxel (Albumin-Bound) 130 mg/m^2, i.v., d1, d8;Carboplatin AUC 5, i.v.,d1;Every 21 days is a cycle, a total of 6 cycles.This study will be divided into three stages.The baseline period:Patients will complete screening tests at baseline to assess eligibility for inclusion criteria.Treatment period:(from the first dose to the last treatment cycle).Imaging tumor assessment was performed every 2 cycles (i.e. 6 weeks).Follow-up period:At the end of the study, patients were followed up by telephone or at the study center every 3 months to collect survival status and subsequent antitumor treatment until death or loss of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age :18-75years old;
2. Histopathological confirmed epithelial ovarian cancer/fallopian tube/peritoneal cancer; Mucinous adenocarcinoma and low-grade serous carcinoma are excluded;
3. Recurrence more than 6 months after the last treatment with taxanes and platinum; Relapse ≤ 3 times; Recovered from the toxicity of the previous chemotherapy to ≤ 1 (hair loss ≤ 2);
4. Relapse confirmed by imaging and CA125:

   1. Clinically evaluable recurrent lesions. According to the RECIST 1.1 , there is at least one measurable lesion as the target lesion. If the target lesion is a lymph node, the shorter diameter is required to be greater than 1.5 cm, and the target lesion has not received radiotherapy;
   2. No clinically evaluable lesions:

   i. Adenocarcinoma cells are confirmed by cytology in the pleural and ascites; ii. Imaging considers that there is tumor recurrence, but the lesions do not meet the measurable standard. They are all small lesions (longest diameter <10 mm or pathological lymph node short diameter ≥10 mm to <15 mm). CA125 ≥ normal upper limit (ULN) 2 times, and CA125 is still showing an upward trend after rechecking after 1 week; c) Patients with recurrence can receive a second cytoreductive surgery. Postoperative R0 resection or residual tumor can be included in the group.
5. ECOG score 0-1;
6. Expected survival time ≥ 3 months;
7. Laboratory tests: absolute neutrophil count (ANC): ≥1.5×10^9/L； platelets (PLT)：≥100×10^9/L；hemoglobin (Hb): ≥90g/L (blood transfusions are allowed to meet or maintain the targets);
8. Liver and renal function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤ULN 2.5times, or <ULN 5times in the presence of liver metastasis; total bilirubin (TBil) level≤ ULN 1.5 times or ≤ ULN 2.5 times when the patients have Gilbert's syndrome; Serum creatinine ≤ ULN 1.5 times or Calculated creatinine clearance ≥ 50 mL/min;
9. Must agree to use effective contraception during the trial; Women of childbearing potential must have a negative serum or urine pregnancy test; Non-lactating patients.
10. Signed the informed consent.

Exclusion Criteria:

1. Patients who had previously received paclitaxel (albumin-bound);
2. Patients who have received abdominal or pelvic radiotherapy;
3. Patients with central nervous system disease or brain metastases;
4. Other malignancies have occurred within the last 5 years, except for cured cervical carcinoma in situ, cutaneous squamous cell carcinoma or controlled basal cell carcinoma of the skin;
5. Prior Grade ≥ 2 sensory or motor neuropathy;
6. Uncontrolled serious medical conditions that, in the opinion of the investigator, would affect the ability of the subject to receive the study regimen, such as concomitant serious medical conditions, including severe heart disease, cerebrovascular disease, uncontrolled diabetes mellitus, uncontrolled hypertension, uncontrolled infection, active peptic ulcer, etc.
7. Allergies to chemotherapeutic drugs or their excipients or intolerant patients;
8. Receive other anti-tumor drugs or participate in other anti-cancer treatment clinical studies within 4 weeks of the first chemotherapy administration;
9. Severe infections occurred within 4 weeks before treatment, including but not limited to infectious complications requiring hospitalization, bacteremia, or severe pneumonia;
10. Human immunodeficiency virus (HIV) positive;
11. Hepatitis B surface antigen (HBsAg) positive. For patients with previous HBV infection or HBV infection cured (the HBsAg is negative, but the total hepatitis B virus core antibody [HBcAb] is positive), if HBV DNA is negative or Undetectable, they can participate in this research;
12. Hepatitis C virus (HCV) antibody positive; Or human immunodeficiency virus and HCV RNA test both positive;
13. Researchers think it is not suitable for enrolling.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-12-09 (Estimated); Primary Completion 2024-02-23 (Estimated); Study Completion 2024-02-23 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | up to 36 months
  From date of randomization until the date of first documented progression or died

SECONDARY OUTCOMES:
Objective response rate(ORR) | up to 36 months
  The proportion of patients with tumor shrinkage reaching a certain amount and for a certain period of time, including cases of CR PR.
Overall survival(OS) | up to 36 months
  From date of randomization until the date of death from any cause
disease control rate(DCR) | up to 36 months
  including CR, PR, SD
hematological toxicity and non-hematological toxicity | up to 36 months
  including hematological toxicity and non-hematological toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Lingying Wu, Study Chair — Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center/ National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China